CLINICAL TRIAL: NCT00462553
Title: A Phase I Study of Sunitinib Malate and Standard Infusion Gemcitabine in Solid Tumors
Brief Title: Sunitinib and Gemcitabine in Treating Patients With Pancreatic Cancer or Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00212; NCI-2009-00212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000539459; CASE 3206; CASE 3206 (Other: Case Western Reserve University); 7731 (Other: CTEP); U01CA062502 (NIH)
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-04

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Sunitinib; Gemcitabine

ARMS (1):
- Arm I (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 OR on days 1, 8, and 15. Patients also receive oral sunitinib malate once daily on days 1-21 OR days 1-28. Treatment repeats every 21 days OR every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar

SUMMARY:
This phase I trial is studying the side effects and best dose of sunitinib and gemcitabine in treating patients with pancreatic cancer or other solid tumors. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in hemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sunitinib together with gemcitabine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of sunitinib malate and gemcitabine hydrochloride in patients with adenocarcinoma of the pancreas or other solid tumors.

II. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 OR on days 1, 8, and 15. Patients also receive oral sunitinib malate once daily on days 1-21 OR days 1-28. Treatment repeats every 21 days OR every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride and sunitinib malate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 10 patients may be treated at the recommended phase II dose (RPTD), which is generally the dose level below the maximally administered dose.

After completion of study treatment, patients are followed for 30 days and then periodically thereafter.

ELIGIBILITY:
Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma OR other solid tumor:

  * Not amenable to curative therapy
  * Previously untreated metastatic pancreatic adenocarcinoma allowed
* Measurable or evaluable disease
* No history of or known brain metastases, spinal cord compression, carcinomatous meningitis, or new evidence of brain or leptomeningeal disease on screening CT scan or MRI scan
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy >= 12 weeks
* Absolute neutrophil count >= 1,500/mm3
* Platelet count >= 100,000/mm3
* Hemoglobin >= 8.5 g/dL
* Bilirubin =< 1.5 mg/dL
* Creatinine normal OR creatinine clearance >= 60 mL/min
* AST and ALT =< 2.5 times upper limit of normal (ULN) (=< 5 times ULN if due to underlying disease)
* Calcium =< 12.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after completion of study therapy
* LVEF normal by MUGA scan or ECHO at baseline
* Deep venous thrombosis or pulmonary embolism allowed provided they are clinically stable and adequately treated
* No preexisting thyroid abnormality that results in the inability to maintain thyroid function in the normal range while using medication
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sunitinib malate
* No history of any of the following within the past 6 months:

  * Myocardial infarction
  * Ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation >= 3 beats in a row)
  * Severe/unstable angina
  * Severe peripheral vascular disease (i.e., claudication)
  * Procedure on peripheral vasculature
  * Coronary/peripheral artery bypass graft
  * Cerebrovascular accident
* No history of any of the following within the past 6 months:

  * Transient ischemic attack;
  * Clinically significant bleeding requiring red blood cell transfusion
* No NYHA class III or IV heart disease:

  * Patients with NYHA class II disease who are stable and on medication are eligible
* No ongoing cardiac dysrhythmias >= grade 2, atrial fibrillation of any grade, or any significant EKG abnormalities
* No hypertension that cannot be controlled by medications to a systolic blood pressure (BP) of < 140 mm Hg and diastolic BP of < 90 mm Hg
* No condition that impairs the ability to swallow and retain sunitinib malate tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No gastrointestinal perforation or intra-abdominal abscess within the past 28 days
* No serious nonhealing infection or bone fracture
* No other severe acute or chronic medical condition, psychiatric condition, or laboratory abnormality that would preclude study therapy
* May have received any number of prior systemic therapies
* More than 4 weeks since prior radiotherapy or surgery and recovered
* More than 4 weeks since other prior therapies and recovered
* Prior gemcitabine hydrochloride allowed
* No prior sunitinib malate or other therapy directed against VEGF, including any of the following:

Sorafenib; Bevacizumab; Vatalanib; AZD2171; VEGF Trap; Investigational antiangiogenic therapy

* More than 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Ketoconazole
  * Itraconazole
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * Indinavir
  * Ritonavir
  * Nelfinavir
  * Saquinavir
  * Atazanavir
  * Delavirdine
* More than 12 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Hypericum perforatum (St. John's wort)
  * Efavirenz
  * Tipranavir
* No concurrent agents with proarrhythmic potential, including any of the following:

  * Terfenadine
  * Quinidine
  * Procainamide
  * Disopyramide
  * Sotalol
  * Probucol
  * Bepridil
  * Haloperidol
  * Risperidone
  * Indapamide
  * Flecainide
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent treatment on another clinical trial:

Participation in non-therapeutic clinical trials allowed

* QTc < 500 msec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events | 28 days

SECONDARY OUTCOMES:
Response rate assessed by Response Evaluation Criteria for Solid Tumors (RECIST) | Up to 3 years
Overall survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Krishnamurthi, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States